CLINICAL TRIAL: NCT01574664
Title: A Prospective, Single-Arm, Multicenter Clinical Study to Evaluate the Safety and Performance of the Health Beacons Radiofrequency Identification (RFID) Localization System for Marking and Retrieving Non-Palpable Breast Lesions
Brief Title: Evaluation of RFID Localization System for Marking and Retrieving Breast Lesions
Status: Withdrawn | Type: Observational
Why Stopped: Not required to be registered
Sponsor: Health Beacons (Industry)
Responsible Party: Sponsor
Other Study IDs: S10-001
Record Dates: First submitted 2012-04-03; First posted 2012-04-10 (Estimated); Last update posted 2020-05-21 (Actual); Status verified 2020-05

CONDITIONS: Non-palpable Breast Lesions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Subjects scheduled to undergo lumpectomy
  Interventions: Device: RFID Tag (Health Beacon)

INTERVENTIONS:
Device: RFID Tag (Health Beacon) — The radiologist or surgeon will place the Health Beacons RFID Tag under ultrasonic or stereotactic guidance. The surgeon will use the Tagfinder to locate the lesion.

SUMMARY:
The goal of this investigation is to obtain clinical data to show the Health Beacons Radiofrequency Identification (RFID) Localization System is safe and performs as intended as a localization device for marking and retrieving a non-palpable surgical target from the breast.

ELIGIBILITY:
Inclusion Criteria:

* Have had stereotactic or ultrasound-guided biopsy with marker placement
* Have a lesion or biopsy marker that is visible under ultrasound
* Have surgical target < 6 cm from the skin when lying supine
* Have a discreet surgical target
* Have a lesion in which the center/focal area is defined
* Be at least 18 years of age or older

Exclusion Criteria:

* Have a palpable lesion that does not require localization
* Require more than one localization needle for localization of the surgical target
* Have undergone previous open surgical biopsy or lumpectomy in the operative breast
* Have an implant in the operative breast
* Have a cardiac pacemaker or defibrillator device

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Female patients
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2017-03 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
The surgical target is visualized in the removed specimen AND the RFID Tag was removed from the patient's breast. | Within 96 hours after lumpectomy
  The study endpoints are known soon after the lumpectomy procedure by 1) confirmation of the pathology lab examination; and 2) retrieval of the implanted RFID tag.

CONTACTS AND LOCATIONS:
Overall Officials: Murray Reicher, MD, Study Director — Health Beacons
Locations (3):
- United States (3):
  - Sharp Memorial Hospital, San Diego, California
  - Harbor-UCLA Medical Center, Torrance, California
  - Exempla Healthcare, Denver, Colorado